CLINICAL TRIAL: NCT06397274
Title: A Phase II, Randomized, Double-Blind, Placebo-controlled, Single-Center Study to Evaluate the Safety and Efficacy of Stemchymal (Allogeneic Adipose-derived Mesenchymal Stem Cells) Infusion for the Treatment of PolyQ Spinocerebellar Ataxia
Brief Title: Stemchymal® for Polyglutamine Spinocerebellar Ataxia
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Steminent US, Inc. (Industry)
Responsible Party: Sponsor
Organization: Steminent Biotherapeutics Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IB02-US
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Spinocerebellar Ataxias
MeSH Terms: conditions — Spinocerebellar Ataxias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Stemchymal® (Experimental)
  Interventions: Biological: Stemchymal
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Stemchymal — Patients will receive Stemchymal® through intravenous infusion
  Arms: Stemchymal®
Biological: Placebo — Patients will receive Placebo through intravenous infusion
  Arms: Placebo

SUMMARY:
The purpose of the clinical trial is to study the therapeutic efficacy and safety of Stemchymal® infusions for polyglutamine spinocerebellar ataxia treatment by a randomized, double-blind, placebo-controlled study design. Eligible subjects will receive Stemchymal® through intravenous infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects are with genotypically confirmed SCA3.
2. Subjects' SARA scores are in the range of 5 to15.
3. Subjects are between 20 and 70 years of age.
4. Subjects who have signed informed consent.
5. Female subjects of child-bearing potential who are capable of conception must be post-menopausal (one year or greater without menses), surgically incapable of childbearing, or practicing effective methods of birth control.
6. Male subjects must be practicing a medically accepted form of contraception during the study period. Abstinence is an acceptable method of contraception.

Exclusion Criteria:

1. Subjects who have been enrolled in any kind of cell therapy within six months prior to screening visit (Visit 1).
2. Female subjects who have a positive pregnancy test result.
3. Subjects who have had severe vital organ diseases, including but not limited to cardiac (e.g., heart failure), liver (e.g., acute hepatic failure or chronic liver cirrhosis), lung (e.g., respiratory failure) and renal (e.g., hemodialysis or peritoneal dialysis) diseases, within six months prior to screening visit (Visit 1).
4. Subjects with immunological disorders (e.g., systemic lupus erythematosus), within six months prior to screening visit (Visit 1).
5. Subjects with other neurological disorders (e.g., Alzheimer's disease), within six months prior to screening visit (Visit 1).
6. Subjects who had received chemotherapy/radiotherapy within five years prior to screening visit (Visit 1).
7. Subjects with any history of malignant tumors.
8. Subjects with dementia or other psychiatric illnesses, including but not limited to disabling depression, bipolar disorder, schizophrenia.
9. Subjects with a Beck Depression Inventory Second Edition (BDI-II) score of over 20 points.
10. Subjects not suitable for this clinical trial according to investigator's judgment.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Change of Scale for the Assessment and Rating of Ataxia (SARA) scores from baseline (week 0) at 6 months (week 24). | 6 months